CLINICAL TRIAL: NCT04280861
Title: Multicomponent Intervention in Caregivers on Quality of Life of People With Dementia: a Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Hospitalari de Vic (Other)
Responsible Party: Principal Investigator, Dr. Pere Roura-Poch, Head of Epidemiology, Consorci Hospitalari de Vic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC278
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease; Caregivers; Quality of Life
MeSH Terms: conditions — Alzheimer Disease | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will participate in multicomponent intervention conducted by and expert psychologist that target different aspects of the caregiving experience (affective responses, communication skills, burden experience, social support and loneliness, cognitive performance, the practice of mindfulness and health-related behaviours). The number of sessions will be 8, 1 session of 90 minutes a week, and the number of participants will be 12-14 per group. In some sessions other collaborators will be invited to participate (social workers, physiotherapist).
  Interventions: Other: Multicomponent Intervention
- Control Group (No Intervention): Usual clinical care,

INTERVENTIONS:
Other: Multicomponent Intervention — Multicomponent intervention conducted by and expert psychologist that target different aspects of the caregiving experience (affective responses, communication skills, burden experience, social support and loneliness, cognitive performance, the practice of mindfulness and health-related behaviours). The number of sessions will be 8, 1 session of 90 minutes a week, and the number of participants will be 12-14 per group. In some sessions other collaborators will be invited to participate (social workers, physiotherapist).
  Other Names: Psychological intervention
  Arms: Intervention Group

SUMMARY:
The main objective is to determine the effectiveness of a multicomponent intervention for caregivers, conducted by an expert psychologist to improve the quality of life of the people with Alzheimer's disease. Secondarily, will be analyzed the effectiveness of this program on improving anxiety and depressive symptoms, burden, happiness, social support and cognitive performance of the caregivers and alleviate the behavioural and psychological symptoms of dementia (BPSD). The investigators analyze the caregiver's and patient's personality as a possible moderator between dependent and independent variables, and the resources utilization before and after intervention.

Methods: randomized study with parallel assignment in two groups: control and intervention group, six-month follow-up. The eligible participants will be 94 adult (≥18 years) caregivers of patients with Alzheimer's disease who follow-up by Osona Integrated Geriatric Unite (Catalonia, Spain).

The intervention group will receive a multicomponent intervention that includes dementia psychoeducation and management, emotional and communication skills, mindfulness and healthy lifestyle. The control group will follow the standard management according to the primary and specialized care professionals' team.

Main measurements: quality of life of the patients at baseline, after intervention and at six-month follow-up through QoL-AD. Secondary measures: they will be determined, at baseline, after the intervention and at six-month follow-up: depression (HDRS) and anxiety (HARS), burden (CBI), happiness (OHQ), quality of life (QoL-AD), social support (UCLA and DUKE-ANC), cognitive performance (neuropsychological assessment) of the caregivers, resources utilization (RUD), BPSD (NPI), cognitive status (MMSE), functional status (IADL) of the patients. Caregiver's personality at baseline and six-month follow-up and dementia characteristics at baseline will be measured. Other measures: sociodemographic and health characteristics of the caregivers and patients.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years of age)
* main caregivers of people with early or mild Alzheimer's disease
* follow-up by Osona Integrated Geriatric Unite (Catalonia)
* signed informed consent.

Exclusion Criteria:

* non stable medical condition the last six months (or any acute or chronic condition that would limit the ability of the patient to participate in the study)
* cognitive impairment (MMSE<24)
* substance abuse
* active psychotherapy
* refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life of the patients after intervention and 6 months follow-up in control and intervention group: Quality of Life-Alzheimer's Disease (QoL-AD) | Baseline, immediately after the intervention and 6 month follow-up
  Quality of life assessed using Quality of Life-Alzheimer's Disease (QoL-AD). The total score ranges from 13 to 52, with a higher number indicating better quality of life

SECONDARY OUTCOMES:
Changes in quality of life of the caregivers: Quality of Life-Alzheimer's Disease (QoL-AD) | Baseline, immediately after the intervention and 6 month follow-up
  Quality of life assessed using Quality of Life-Alzheimer's Disease (QoL-AD). The total score ranges from 13 to 52, with a higher number indicating better quality of life
Changes in loneliness | Baseline, immediately after the intervention and 6 month follow-up
  UCLA - University of California Loneliness Scale. The total score ranges from 10 to 40. Score: 20-30: moderate depression, and ≥ 20: severe loneliness
Changes in depression of the caregivers | Baseline, immediately after the intervention and 6 month follow-up
  HDRS: Hamilton Depression Rating Scale. Score: 0-7: No depression; 8-13: Mild depression; 14-18: Moderate depression; 19-22: Severe depression and ≥ 23: Very severe depression
Characteristics and changes in caregivers personality | Baseline, immediately after the intervention and 6 month follow-up
  NEO-Personality Inventory-R. For each scale, the interval 20-35 indicates very low scores. The interval 35-45 indicates low scores. The interval 45-55 indicates average scores. The interval 55-65 indicates high scores. The interval 65-80 indicates very high scores.
Changes in cognitive performance of the caregivers | Baseline, immediately after the intervention and 6 month follow-up
  Neuropsychological assessment
Changes in sleep patterns of the caregivers | Baseline, immediately after the intervention and 6 month follow-up
  PSQI: Pittsburgh Sleep Quality Index. The total score ranges from 0 to 21, with a higher number indicating better sleep quality
Changes of the resource utilization | Baseline, immediately after the intervention and 6 month follow-up
  RUD: Resource Utilization in Dementia Questionnaire Scale
Changes in cognitive status of the patients | Baseline, immediately after the intervention and 6 month follow-up
  MMSE (Mini Mental State Examination). Range scores 0 to 30. Score: 24-30: no cognitive impairment; 19-23: mild cognitive impairment; 10-18: moderate cognitive impairment; ≤9: severe cognitive impairment
Changes in Behavioural and Psychological Symptoms of Dementia | Baseline, immediately after the intervention and 6 month follow-up
  NeuroPsychiatric Inventory. 12 scales, the domain total score is the product of the frequency score multiplied by the severity score for that behavioral domain
Satisfaction with the intervention: Interview | Immediately after the intervention
  Satisfaction Interview
Changes in perceived social support of the caregivers | Baseline, immediately after the intervention and 6 month follow-up
  DUKE-ANC. The total score ranges from 11 to 55, with a higher number indicating worse perceibed social support
Anxiety | Baseline, immediately after the intervention and 6 month follow-up
  HARS- Hamilton Anxiety Rating Scale. Score: 0-5: No anxiety; 6-14: Mild anxiety; ≥ 15: Moderate to severe anxiety
Happiness | Baseline, immediately after the intervention and 6 month follow-up
  OHQ : Oxford Happiness Questionnaire. The total score ranges from 8 to 54, with a higher number indicating better subjective wellness
Burden in caregivers | Baseline, immediately after the intervention and 6 month follow-up
  CBI: Caregiver Burden Interview. Total score ranges from 22 to 110. Score: 22-46: No burden; 47-55: burden; 56-110: intense burden
Functional status of the patients | Baseline, immediately after the intervention and 6 month follow-up
  IADL: Instrumental. Activities of Daily Living. Sum the binary responses of each activity, sum the eight responses The higher the score, the greater the person's abilities

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Hospitalari de Vic, Vic, Barcelona, Spain